CLINICAL TRIAL: NCT02576873
Title: Long-term Outcome of End-stage Renal Disease Patients Treated With High-efficiency Hemodiafiltration: a Historical Cohort of a Single-center in South East Asia
Brief Title: Long-term Outcome of End-stage Renal Disease Patients Treated With Hig-efficiency Hemodiafiltration
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Assistant Professor, Chulalongkorn University
Other Study IDs: 455/56
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: End-stage Renal Disease
Keywords: Survival; Hemodiafiltration; End-stage renal disease; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hemodiafiltration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodiafiltration: End-stage renal disease patients who were treated with high-efficiency hemodiafiltration for more than 6 months
  Interventions: Other: Hemodiafiltration

INTERVENTIONS:
Other: Hemodiafiltration — Hemodiafiltration treatments were prescribed to the patients as their long-term renal replacement therapies

SUMMARY:
A retrospective cohort study was conducted in 66 end-stage renal disease patients who underwent high-efficiency hemodiafiltration technique in King Chulalongkorn Memorial Hospital between 2001-2013 to determine the survival rate as well as other long-term outcome.

DETAILED DESCRIPTION:
Growing evidences suggested the superiority of high-efficiency hemodiafiltration (HDF) which could provide both diffusion and convection in a single therapy compared with the conventional hemodialysis. However, the long-term, upto 10 years, outcome still limited. This retrospective cohort study was conducted in 66 end-stage renal disease patients who underwent high-efficiency hemodiafiltration technique in a single-center, King Chulalongkorn Memorial Hospital, between 2001-2013 to determine the survival rate as well as other long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Be diagnosed end-stage renal disease for more than one year
* Have been regularly received long-term hemodiafiltration for more than 6 months.

Exclusion Criteria:

* Patients who received hemodiafiltration less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End-stage renal disease patients who had been received long-term hemodiafiltration at King Chulalongkorn Memorial hospital during 2001-2013
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Survival rate | 10 years
  The Kaplan-Meier survival curve and mean survival time will be demonstrated for primary outcome.

SECONDARY OUTCOMES:
Comparison of survival differences between patients who start renal replacement therapy with HDF and who switched from hemodialysis as well as between diabetic and non-diabetic patient. | 10 years
  Survival differences between groups will be evaluated with the Kaplan-Meier method and compared using the log-rank test. The comparative groups include:
  * Patient who start renal replacement therapy with HDF (incident cases) vs. who switched from hemodialysis (prevalence cases)
  * Diabetic vs. Non-diabetic patients
Factors that associated with all-cause mortality | 10 years
  univariate and multivariate analysis the factors that might affected the long-term outcomes. The factors include dialytic parameters (spKt/Vurea, TAC urea), nutritional parameters (nPNA, albumin), inflammatory parameter (hsCRP), and biochemical parameters (BUN, Cr, Ca, Phosphate, iPTH, beta2-microglobulin, Hb, Ferritin, Transferrin saturation, Cholesterol, Triglyceride, HDL, and LDL)

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Pathumwan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No